CLINICAL TRIAL: NCT02956161
Title: Effects of Synchronised Auditory Stimulations of the Sleep Slow Oscillation on Deep Sleep
Brief Title: Effects of Synchronised Auditory Stimulations of the Sleep Slow Oscillation on Deep Sleep Quality
Acronym: STIMENPHASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dreem (Industry)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STIMENPHASE
Record Dates: First submitted 2016-10-20; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Sleep; Auditory stimulations; Slow oscillations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Up phase stimulation (Experimental): Auditory stimulations are delivered in synchrony with the up phase of slow oscillations during N3 sleep stage.
  Interventions: Device: Stimulation of up-phase of sleep slow oscillation
- Random phase stimulation (Experimental): Auditory stimulations are randomly delivered during N3 sleep stage.
  Interventions: Device: Random stimulation of up phase of sleep slow oscillation
- No stimulation (Sham Comparator): The device is worn without any auditory stimulations delivered.
  Interventions: Device: No stimulation

INTERVENTIONS:
Device: Stimulation of up-phase of sleep slow oscillation
  Arms: Up phase stimulation
Device: Random stimulation of up phase of sleep slow oscillation
  Arms: Random phase stimulation
Device: No stimulation
  Arms: No stimulation

SUMMARY:
This monocentric, cross-over, randomised, double blind and placebo-controlled study evaluates the effects of auditory stimulations of the sleep slow oscillation on deep sleep quality.

DETAILED DESCRIPTION:
Sleep quality impairment has long been identified as a risk factor to develop cardio-vascular, metabolic and more recently neurodegenerative diseases. The slow wave sleep, characterized by slow oscillations, has a major role on memory and hormones releasing. Here, we aim to assess a miniaturized sleep device that would automatically detect and stimulate sleep slow oscillations with sounds to enhance deep sleep quality.

The subjects realize 3 conditions :

* Up condition : Auditory stimulations are delivered in synchrony with the up phase of slow oscillations during N3 sleep stage.
* Random condition : Auditory stimulations are randomly delivered during N3 sleep stage.
* Placebo condition: The device is worn without any auditory stimulations delivered.

The subjects are equipped with a reference polysomnography and the auditory stimulation device during 3 nights and one habituation night prior to them. A wash out period of 6 days between each night will be respected.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject
* moderate morningness, intermediate or moderate eveningness chronotype (Horne & Östberg questionnaire)

Exclusion Criteria:

* sleep disorder according to the ICSD-3 or DSM-5
* travelling away from more than a time zone in the previous month
* acute or chronic disorders (cardio-vascular, respiratory, neurologic, psychiatric)
* night shifts work
* smoking more than 5 cigarettes per day
* drinking more than 5 glass of alcohol per week
* consuming excessive drinks with xanthics (coffee, tea, coke more than 6 cups per day).
* having a body mass index >30kg.m -2
* being pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Variation of the amplitude of sleep slow oscillations | 3 days
  Amplitude of sleep slow oscillation assessed during N3 sleep stages throughout 3 separate nights. The analysis is based on electroencephalography signal.

SECONDARY OUTCOMES:
Variation of the number of sleep slow oscillations | 3 days
  Number of sleep slow oscillation assessed during N3 sleep stages throughout 3 separate nights. The analysis is based on electroencephalography signal.
Variation of N3 sleep stage duration | 3 days
  N3 sleep duration assessed throughout 3 separate nights. The analysis is based on double scoring of polysomnography signal.
Variation of the number of remembered words in declarative memory tasks (word pair task) | 3 days
  Number of remembered words assessed 3 separate days (30 min after awakening).
Variation of mood assessment measured with the profile of mood scale (POMS) | 3 days
  Mood assessed 3 separate days (30 min after awakening).
Variation of subjective sleepiness measured with the Karolinska sleepiness scale (KSS) | 3 days
  Subjective sleepiness assessed 3 separate days (30 min after awakening).
Variation of average response time variation and omissions in the Psychomotor vigilance task (PVT) | 3 days
  Psychomotor vigilance assessed 3 separate days (30 min after awakening).
Variation of salivary cortisol concentration | 3 days
  Salivary cortisol concentration assessed 3 separate days (5 min after awakening).
Variation of salivary testosterone concentration | 3 days
  Salivary testosterone concentration assessed 3 separate days (5 min after awakening).
Variation of mental rotation capacity (mental rotatory task) | 3 days
  Mental rotation capacity assessed 3 separate days (30 min after awakening).

CONTACTS AND LOCATIONS:
Overall Officials: Damien Léger, MD, PhD, Principal Investigator — EA 7330 VIFASOM, University of Paris Descartes, Sorbonne Cité, Paris; Mounir Chennaoui, PhD, Study Director — EA 7330 VIFASOM, University of Paris Descartes, Sorbonne Cité, Paris
Locations (1):
- Centre du Sommeil et de la Vigilance, Hotel-Dieu de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Yes